CLINICAL TRIAL: NCT00446771
Title: A Pharmacokinetic and Bioavailability Study of Mannitol for Inhalation Using Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syntara (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DPM-PK-101
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Mannitol

INTERVENTIONS:
Drug: Mannitol

SUMMARY:
The study has an open-label, randomized, crossover design, in which each subject will receive mannitol powder for inhalation using a dry powder inhaler with and without premedication with a bronchodilator, mannitol powder for inhalation in capsules administered orally, and mannitol in a commercial formulation designed for intravenous use.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed a written informed consent form.
* Subject is a normal male volunteer between 18 and 65 years of age.
* Subject is willing to comply with the procedures of the study and to remain in the clinical unit for the scheduled visits.
* Subject is willing to abstain from chewing gum for the duration of the study.

Exclusion Criteria:

* Subject has asthma or other disease affecting the lungs or airways.
* Subject has a history indicating possible airway hyperresponsiveness.
* Subject is allergic to mannitol or gelatin or a known intolerance to intravenous mannitol.
* Subject uses inhaled drugs (legal or illegal).
* Subject uses oral bronchodilator drugs.
* Subject has celiac disease, Crohn's disease or other disease affecting intestinal absorption.
* Subject has renal impairment or other condition that would affect urine collection.
* Subject's weight deviates by more than 15% from the ideal weight listed for his height in the Metropolitan Life table.
* Subject is a smoker.
* Subject has participated in another clinical trial within the past 30 days.
* Subject has used chewing gum within the past 72 hours.
* Subject needs to use bisphosphonates, non-steroidal anti-inflammatory agents, or other drugs known to affect intestinal permeability on a chronic basis.
* Subject has used non-steroidal anti-inflammatory agents within the past 72 hours

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2006-10; Study Completion 2006-11

PRIMARY OUTCOMES:
To determine the absolute bioavailability of mannitol powder for inhalation by comparison to mannitol administered intravenously.
To determine the relative bioavailability of mannitol powder for inhalation by comparison to orally administered mannitol.
To determine the pharmacokinetic parameters of systemically available mannitol after administration of mannitol powder by inhalation.

SECONDARY OUTCOMES:
A secondary objective of the study is to provide information on the urinary excretion of mannitol after each of the routes of administration.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Humberstone, Principal Investigator — Nucleus Networks